CLINICAL TRIAL: NCT01612013
Title: Intravenous High Dose of N-acetylcysteine and Sodium Bicarbonate for the Prevention of Contrast-induced Acute Injury: a Randomized Controlled Trial
Brief Title: Intravenous High Dose NAC and Sodium Bicarbonate for the Prevention of Contrast-induced Acute Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Hospital das Forças Armadas, Brazil (Other); InCor Heart Institute (Other)
Responsible Party: Principal Investigator, Antonio Jose de Almeida Inda Filho, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EPM1FU311281
Record Dates: First submitted 2012-05-30; First posted 2012-06-05 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Acute Renal Failure
Keywords: N-acetylcysteine; angiography; contrast medium; contrast-induced nephropathy; sodium bicarbonate
MeSH Terms: conditions — Acute Kidney Injury | interventions — Sodium Bicarbonate; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Intravenous NAC plus saline (Active Comparator): Acetylcysteine was given via intravenous bolus at a rate of 150 mg/kg over 60 min immediately before contrast exposure and followed by 50 mg/kg during and for 6 hours after the procedure. Saline (0.9 percent) was given intravenous at a rate of 1 ml/Kg/h over 60 min prior and followed at the same rate during and for the next 6 hours the procedure.
  Interventions: Drug: Intravenous NAC plus saline; Drug: NAC plus saline
- Sodium bicarbonate plus saline (Active Comparator): Sodium bicarbonate solution (Sodium bicarbonate 8.4%, Equiplex, Brazil) was given by adding fifteen ampoules of sodium bicarbonate (150 mEq of sodium) to 1 L of 5% dextrose. Infusion in bolus began 60 min prior to the start of contrast administration at 3.5 ml/Kg/h, decreased to 1.18 ml/Kg/h during the contrast exposure and for the next 6 hours after the procedure. Saline (0.9 percent) was given IV at a rate of 1 ml/Kg/h over 60 min prior to the start of contrast administration and followed at the same rate during and for the next 6 hours after the procedure.
  Interventions: Drug: Sodium bicarbonate plus saline
- NAC plus sodium bicarbonate plus saline (Active Comparator): Acetylcysteine was given intravenous at a rate of 150 mg/kg over 60 min before contrast exposure and followed by 50 mg/kg during and for 6 hours after the procedure. Sodium bicarbonate solution (150 mEq/L of sodium) was given in bolus began 60 min before contrast administration at 3.5 ml/Kg/h, decreased to 1.18 ml/Kg/h during and for the next 6 hours of the procedure. Saline was given intravenous at a rate of 1 ml/Kg/h over 60 min prior to the start of contrast administration and followed at the same rate during and for the next 6 hours after the procedure.
  Interventions: Drug: NAC plus sodium bicarbonate plus saline
- Saline (Placebo Comparator): Saline (0.9 percent) was given IV at a rate of 1 ml/Kg/h over 60 min prior to the start of contrast administration and followed at the same rate during and for the next 6 hours after the procedure.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Sodium bicarbonate plus saline — Sodium bicarbonate solution (Sodium bicarbonate 8.4%, Equiplex, Brazil) was given by adding fifteen ampoules of sodium bicarbonate (150 mEq of sodium) to 1 L of 5% dextrose. Infusion in bolus began 60 min prior to the start of contrast administration at 3.5 ml/Kg/h, decreased to 1.18 ml/Kg/h during the contrast exposure and for the next 6 hours after the procedure. Saline (0.9 percent) was given IV at a rate of 1 ml/Kg/h over 60 min prior to the start of contrast administration and followed at the same rate during and for the next 6 hours after the procedure.
  Arms: Sodium bicarbonate plus saline
Drug: Intravenous NAC plus saline — Acetylcysteine (Flucistein 100 mg/ml, Neo Química, Brazil) was given via IV bolus at a rate of 150 mg/kg in 500 ml dextrose 5% over 60 min immediately before contrast exposure and followed by 50 mg/kg in 500 ml dextrose 5% during the contrast exposure and for 6 hours after the procedure. Saline (0.9 percent) was given IV at a rate of 1 ml/Kg/h over 60 min prior to the start of contrast administration and followed at the same rate during and for the next 6 hours after the procedure.
  Arms: Intravenous NAC plus saline
Drug: NAC plus sodium bicarbonate plus saline — Acetylcysteine was given intravenous at a rate of 150 mg/kg over 60 min before contrast exposure and followed by 50 mg/kg during the contrast exposure and for 6 hours after the procedure. Sodium bicarbonate solution(150 mEq of sodium) was began 60 min prior to the start of contrast administration at 3.5 ml/Kg/h, decreased to 1.18 ml/Kg/h during the contrast exposure and for the next 6 hours after the procedure. Saline was given intravenous at a rate of 1 ml/Kg/h over 60 min prior to the start of contrast administration and followed at the same rate during and for the next 6 hours after the procedure.
  Arms: NAC plus sodium bicarbonate plus saline
Drug: Saline — Saline (0.9 percent) was given IV at a rate of 1 ml/Kg/h over 60 min prior to the start of contrast administration and followed at the same rate during and for the next 6 hours after the procedure.
  Arms: Saline
Drug: NAC plus saline — Acetylcysteine was given via intravenous bolus at a rate of 150 mg/kg over 60 min immediately before contrast exposure and followed by 50 mg/kg during and for 6 hours after the procedure. Saline (0.9 percent) was given intravenous at a rate of 1 ml/Kg/h over 60 min prior and followed at the same rate during and for the next 6 hours the procedure.
  Arms: Intravenous NAC plus saline
Drug: NAC plus sodium bicarbonate plus saline — Acetylcysteine was given intravenous at a rate of 150 mg/kg over 60 min before contrast exposure and followed by 50 mg/kg during and for 6 hours after the procedure. Sodium bicarbonate solution (150 mEq/L of sodium) was given in bolus began 60 min before contrast administration at 3.5 ml/Kg/h, decreased to 1.18 ml/Kg/h during and for the next 6 hours of the procedure. Saline was given intravenous at a rate of 1 ml/Kg/h over 60 min prior to the start of contrast administration and followed at the same rate during and for the next 6 hours after the procedure.
  Arms: NAC plus sodium bicarbonate plus saline

SUMMARY:
Contrast-induced acute kidney injury is a common cause of acquired in-hospital renal insufficiency and is associated with prolonged hospitalization and unfavorable early and late outcomes. The investigators sought to compare 4 different strategies (intravenous high-dose of N-acetylcysteine, sodium bicarbonate, the combination of both, and saline alone) in the prevention of contrast-induced acute kidney injury in patients undergoing coronary angiography using high-osmolar contrast media defined by creatinine and cystatin C serum levels.

ELIGIBILITY:
Inclusion Criteria:

* eligible patients include individuals aged 18 year or older with normal renal function who were schedule to undergo cardiac catheterization. During the randomized study, consecutive eligible patients schedule for exposure to the ionic, high osmolality (2130 mOsm/Kg) contrast agent Ioxitalamato.

Exclusion Criteria:

* using metformin or nonsteroidal antiinflammatory drugs within the previous 48 hours
* intake of nephrotoxic drugs during the previous seven days
* pregnancy
* lactation
* intravascular administration of an iodinated contrast medium within the previous two days
* emergency catheterization
* pulmonary edema
* acutely decompensate congestive heart failure
* history of serious reactions to iodinated contrast mediums
* renal transplantation
* end-stage renal disease necessitating dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2005-05; Primary Completion 2009-05 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The development of contrast-induced acute kidney injury based either on the creatinine and/or Cystatin C increase between day 0 and 72 hours. | 72 hours
  The primary end point of the study was the development of contrast-induced acute kidney injury based either on the creatinine and/or Cystatin C increase between day 0 (when contrast media was administered) and 72 hours (creatinine; Cystatin C increase ≥ 0.3 mg/dL increase and/or 10% increase, respectively within 72 hours after contrast media administration).

SECONDARY OUTCOMES:
The secondary end point was development of CI-AKI in a subgroup of high-risk patients, including patients with diabetes mellitus and those with pre-existent kidney disease defined as calculated creatinine clearance < 60 ml/min/1.73m2. | 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Forcas Armadas - Fundacao Zerbine - INCOR, Brasília, Federal District, Brazil

REFERENCES:
- [Derived] Inda-Filho AJ, Caixeta A, Manggini M, Schor N. Do intravenous N-acetylcysteine and sodium bicarbonate prevent high osmolal contrast-induced acute kidney injury? A randomized controlled trial. PLoS One. 2014 Sep 25;9(9):e107602. doi: 10.1371/journal.pone.0107602. eCollection 2014. PMID 25254489